CLINICAL TRIAL: NCT02632617
Title: coRonary assEssment of Preoperative vaLvulopathy pAtients Using ComputEd Tomographic Angiography (REPLACE)
Acronym: REPLACE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: Guangdong Provincial People's Hospital (Other); West China Hospital (Other); Air Force Military Medical University, China (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Bin Lu, Professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2015-681; 2012-XHGX05 (Other Grant/Funding Number: Peking Union Medical College); 2011-XH3 (Other Grant/Funding Number: Peking Union Medical College)
Record Dates: First submitted 2015-12-05; First posted 2015-12-17 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Heart Valve Diseases; Coronary Artery Disease
Keywords: Heart Valve Diseases; Coronary Artery Disease; Computed Tomographic Angiography; Preoperative Procedure
MeSH Terms: conditions — Heart Valve Diseases; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CTA Group: Participants in CTA group will primarily receive computed tomographic angiography examination before surgery. Those with positive findings in CTA (≥50% diameter stenosis in main coronary artery) or uncertain diagnosis caused by motion artifact or calcium artifact are required to undergo ICA, and coronary artery bypass grafting (CABG) is recommended in patients with significant stenosis according to the ICA result. Participants with negative findings in CTA do not need further coronary artery evaluation, and CABG won't be performed during the surgery.
  Interventions: Other: Computed tomographic angiography
- ICA Group: Participants in ICA group will undergo ICA as guideline recommend before surgery, coronary artery bypass grafting (CABG) is recommended in patients with significant stenosis

INTERVENTIONS:
Other: Computed tomographic angiography — Preoperative examination is needed in patients with valvular disease. The invasive coronary angiography is used for patients in ICA group, while the computed tomographic angiography is used as a gatekeeper and invasive coronary angiography is selectively used for patients in CTA group.
  Other Names: CTA
  Groups: CTA Group

SUMMARY:
Preoperative detection of combined coronary artery disease by invasive coronary angiography (ICA) is recommended in American Heart Association (AHA)/American College of Cardiology (ACC) guidelines for most patients (>40 yrs male or postmenopausal female) scheduled for heart valve surgery, but the low incident rate of coronary artery disease implied guidelines for the vast majority who ultimately will not undergo revascularization. Computed tomography angiography (CTA) has emerged as an alternative diagnosis procedure, which has the following advantages: non-invasive, low cost, provide information of lung and mediastinum. Our study is to evaluate the feasibility of computed tomography, instead of conventional invasive coronary angiography in evaluating coronary artery lesion prior to the heart valvular operation.

DETAILED DESCRIPTION:
Valvular heart disease is common in China, either rheumatic or degenerative, and valvular repair or replacement surgery is the important therapeutic method. In all forms of heart valvular disease, combined coronary artery disease worsens perioperative prognosis. Preoperative detection of combined coronary artery disease with invasive coronary angiography is recommended in most patients scheduled for valve surgery, while incidence rate of coronary artery disease in patients with valvular disease showed that only 3%-19% patients were diagnosed with significant stenosis. Although invasive coronary angiography is considered a safe procedure, it still carries a small risk of major (death, stroke, or vascular dissection) and minor (inguinal hematoma) complications. Furthermore, the catheterization procedure is rather expensive, as its invasive nature involves admission to a hospital and requires surveillance by an experienced team. As a non-invasive alternative diagnosis procedure, coronary computed tomographic angiography has showed promising performance with high negative predictive value (95%-100%). Furthermore, computed tomography is a noninvasive procedure with low risk and cost, and it can be easily performed at the clinic. Except for evaluation of coronary artery, computed tomography can also provide information of lung, mediastinum and cardiac structure, which may help physicians make early diagnosis and treatment. Computed tomography is not routinely utilized in clinical practice.

Our study is a prospective multicenter study to assess the feasibility and safety of adding computed tomography as a gatekeeper and perform invasive coronary angiography selectively prior to valvular surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Male ≥ 40 years old; postmenopausal female;
* Patients scheduled to undergo valvular replacement or repair;
* Patients providing written informed consent;

Exclusion Criteria:

* Patients with definite coronary artery disease history (Prior myocardial infarction, percutaneous coronary intervention or CABG);
* Patients with objective evidence of myocardial ischemia;
* Underwent CTA or ICA in 6 months;
* With contraindications to CTA/ICA (allergic to contrast medium, peripheral arterial occlusive disease, chronic kidney disease with estimated glomerular filtration rate (eGFR) less than 15ml/min.1.73m2 )

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population in our study comprise pre-operative individuals with valvular disease who are recommended for ICA by the 2014 ACC/AHA guideline
Sampling Method: Non-Probability Sample
Enrollment: 2644 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-01 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of cardiovascular complications and mortality [Perioperative Safety] | POD 30 days
  Incidence rates of intraoperative and postoperative cardiovascular complications and mortality caused by coronary stenosis within 30 days after the surgery will be compared between the two groups.

SECONDARY OUTCOMES:
Effectiveness of the coronary artery evaluation protocol | 48 hours after coronary evaluation (CTA or ICA)
  Proportion of patients with significant stenosis(stenosis ≥50%)
Effectiveness of the coronary artery evaluation protocol | 24h after the operation
  Proportion of patients underwent expected CABG will be compared.

OTHER OUTCOMES:
Safety of the coronary examination (CTA or ICA) | 24 hours after the examination
  radiation dose, contrast volume and adverse event in 24 hours after the examination
Hospitalization cost of patients | During hospital stay, an average of 10 days
  medical cost during the hospital include examination cost, operation cost, drug cost and other cost

CONTACTS AND LOCATIONS:
Overall Officials: Bin Lu, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (5):
- China (5):
  - Fuwai Hospital, Beijing, Beijing Municipality
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xijing Hospital, Xian, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Meijboom WB, Mollet NR, Van Mieghem CA, Kluin J, Weustink AC, Pugliese F, Vourvouri E, Cademartiri F, Bogers AJ, Krestin GP, de Feyter PJ. Pre-operative computed tomography coronary angiography to detect significant coronary artery disease in patients referred for cardiac valve surgery. J Am Coll Cardiol. 2006 Oct 17;48(8):1658-65. doi: 10.1016/j.jacc.2006.06.054. Epub 2006 Sep 26. PMID 17045904
- [Background] Nishimura RA, Otto CM, Bonow RO, Carabello BA, Erwin JP 3rd, Guyton RA, O'Gara PT, Ruiz CE, Skubas NJ, Sorajja P, Sundt TM 3rd, Thomas JD, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Creager MA, Curtis LH, DeMets D, Guyton RA, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Stevenson WG, Yancy CW; American College of Cardiology; American College of Cardiology/American Heart Association; American Heart Association. 2014 AHA/ACC guideline for the management of patients with valvular heart disease: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Thorac Cardiovasc Surg. 2014 Jul;148(1):e1-e132. doi: 10.1016/j.jtcvs.2014.05.014. Epub 2014 May 9. No abstract available. PMID 24939033
- [Background] Gilard M, Cornily JC, Pennec PY, Joret C, Le Gal G, Mansourati J, Blanc JJ, Boschat J. Accuracy of multislice computed tomography in the preoperative assessment of coronary disease in patients with aortic valve stenosis. J Am Coll Cardiol. 2006 May 16;47(10):2020-4. doi: 10.1016/j.jacc.2005.11.085. Epub 2006 Apr 24. PMID 16697319
- [Background] Yin WH, Lu B, Gao JB, Li PL, Sun K, Wu ZF, Yang WJ, Zhang XQ, Zheng MW, McQuiston AD, Meinel FG, Schoepf UJ. Effect of reduced x-ray tube voltage, low iodine concentration contrast medium, and sinogram-affirmed iterative reconstruction on image quality and radiation dose at coronary CT angiography: results of the prospective multicenter REALISE trial. J Cardiovasc Comput Tomogr. 2015 May-Jun;9(3):215-24. doi: 10.1016/j.jcct.2015.01.010. Epub 2015 Jan 22. PMID 25843243
- [Background] Yin WH, Lu B, Li N, Han L, Hou ZH, Wu RZ, Wu YJ, Niu HX, Jiang SL, Krazinski AW, Ebersberger U, Meinel FG, Schoepf UJ. Iterative reconstruction to preserve image quality and diagnostic accuracy at reduced radiation dose in coronary CT angiography: an intraindividual comparison. JACC Cardiovasc Imaging. 2013 Dec;6(12):1239-49. doi: 10.1016/j.jcmg.2013.08.008. Epub 2013 Oct 23. PMID 24269265